CLINICAL TRIAL: NCT06673134
Title: Prospective Registry Study and Clinical Observation of Children With Crohn's Disease
Brief Title: Prospective Cohort Establishment and Clinical Observation of Children With Crohn's Disease
Acronym: CD
Status: Active, not recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Biao Zou, Attending physician, pediatric department, Tongji Hospital
Other Study IDs: 63639582
Record Dates: First submitted 2024-10-26; First posted 2024-11-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Crohn Disease
Keywords: Corticosteroids; immunosuppressants; biological agents;; Exclusive enteral nutrition;; pediatric
MeSH Terms: conditions — Crohn Disease | interventions — Enteral Nutrition; Nutritional Status; Immunotherapy; macrophage-derived immunosuppressor factor; Biological Factors; Biological Therapy; Glucocorticoids; Fecal Microbiota Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Serum specimen, Stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- enteral nutrition group: enteral nutrition therapy, including exclusive enteral nutrition and Partial enteral nutrition
  Interventions: Drug: Immunotherapy; Drug: biological agents; Drug: Glucocorticoids; Other: fecal microbiota transplantation
- Glucocorticoid group: Glucocorticoid therapy
  Interventions: Drug: enteral nutrition; Drug: biological agents; Other: fecal microbiota transplantation
- Immunosuppressive group: Immunosuppressive therapy
  Interventions: Drug: enteral nutrition; Drug: biological agents; Other: fecal microbiota transplantation
- Fecal Microbiota Transplantation group: Fecal Microbiota Transplantation therapy
  Interventions: Drug: enteral nutrition; Drug: Immunotherapy; Drug: biological agents; Drug: Glucocorticoids
- Biologics group: Biologics therapy, Including various types of biological agents, as well as domestic biological agents (Taizhou Mabtech Pharmaceutical Co.,Ltd).
  Interventions: Drug: enteral nutrition; Drug: Immunotherapy; Drug: Glucocorticoids; Other: fecal microbiota transplantation

INTERVENTIONS:
Drug: enteral nutrition — exclusive enteral nutrition therapy or Partial enteral nutrition
  Other Names: nutrition
  Groups: Biologics group; Fecal Microbiota Transplantation group; Glucocorticoid group; Immunosuppressive group
Drug: Immunotherapy — Immunosuppressants therapy, Including thalidomide, azathioprine, methotrexate, etc
  Other Names: immunosuppressor
  Groups: Biologics group; Fecal Microbiota Transplantation group; enteral nutrition group
Drug: biological agents — Inflixima , domestic infliximab (Taizhou Mabtech Pharmaceutical Co.,Ltd) and Adalimumab , etc
  Other Names: biotherapy
  Groups: Fecal Microbiota Transplantation group; Glucocorticoid group; Immunosuppressive group; enteral nutrition group
Drug: Glucocorticoids — Glucocorticoids treatments are given
  Other Names: glucocorticoid
  Groups: Biologics group; Fecal Microbiota Transplantation group; enteral nutrition group
Other: fecal microbiota transplantation — Fecal bacteria transplantation treatment, transplantation routes include enema, TET route, capsule fecal bacteria route, etc
  Other Names: Flora transplantation
  Groups: Biologics group; Glucocorticoid group; Immunosuppressive group; enteral nutrition group

SUMMARY:
To evaluate the clinical manifestations, treatment options, and improved clinical outcomeof children with Crohn's disease in real-world Settings: (1) analysis of clinical manifestations; (2) probability of using the same treatment options; (3) Clinical outcome;

DETAILED DESCRIPTION:
This study will aim to enroll approximately 100 patients with Crohn Disease (CD). All patients who have CD will be evaluated at the Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology. Patients who are eligible for the study will be identified during these regularly scheduled clinic visits. Patients and guardians who express interest will be set up for a meeting with a clinical research coordinator who will go over the study in detail and will obtain informed consent. Before the therapeutic intervention，stool samples will be checked for ova and parasites, C. difficile toxin and fecal calprotectin (FCP). Serum tests will include erythrocyte sedimentation rate (ESR), C-reactive protein (CRP), Anti-nuclear antibodies (ANA), complete blood cell count, HIV, screening for Hepatitis A, B, C (hep A IgM, hep B surface antigen and antibody, Hep C antibody), and creatinine. Fecal tests included 16S rDNA flora detection and metabolite detection. Patients with CD will undergo colonoscopy, which is considered part of standard of care for patients with ongoing inflammation and is not considered a study procedure.

Dynamic monitoring follow-up up to 102 weeks, dynamic assessment of relevant indicators, such as ESR, CRP, FCP and endoscopy, etc. This study is an observational study, without intervention in the treatment of patients. Patients will accept the treatment plan formulated by the attending physician. Treatment options include: enteral nutrition (EEN/ PEN, reason, route of administration, dose, course of treatment); glucocorticoids (reason, route of administration, dose, course of treatment); immunosuppressants (reason, route of administration, dose, course of treatment); biologics (including domestic infliximab (Taizhou Mabtech Pharmaceutical Co.,Ltd)) (dose, duration, effectiveness, safety, and economy); fecal microbiota transplantation (cause, transplantation routes, capsule fecal transplants, dose, course of treatment); the medical costs and resource consumption of the treatment of Crohn's disease in children. The difference of efficacy of the above treatment schemes was recorded, the treatment outcome was compared, and the transformation of treatment schemes was discussed. Researchers and patients will truthfully register the corresponding data generated by clinical practice from the doctors and patients respectively, collect the laboratory examination and evaluation data of doctors during the visit, and combine the hospital visit and electronic information system. Statistical analysis was performed after follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Children under 17 years old;
* Children with a definite diagnosis of Crohn's disease;
* Patients and their guardians must sign informed consent;

Exclusion Criteria:

* Other conditions deemed inappropriate by the doctor to participate in the study;

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 100
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-07-24 (Estimated); Study Completion 2028-07-24 (Estimated)

PRIMARY OUTCOMES:
To evaluate the clinical manifestations, treatment options, and clinical outcomes of Crohn's disease in children in real-world Settings | 14 weeks
  14 weeks clinical response rate.

SECONDARY OUTCOMES:
Clinical remission of different treatment regimens | 14 and 54 weeks
  Clinical remission rates at 14 and 54 weeks ( Pediatric Crohn's Disease Activity Index (PCDAI)≤10, PCDAI<10.0 was defined as the stage of clinical remission, 10.0~27.5 as the stage of clinical mild activity, 30.0~37.5 as the stage of clinical moderate activity, and 40.0~100.0 as the stage of clinical severe activity.)
Clinical response of different treatment regimens | 54 weeks
  Clinical response rate at 54 weeks (PCDAI reduction ≥15 points and total PCDAI≤30 points)
Endoscopic response of different treatment regimens | 14 and 54 weeks
  Endoscopic response rate at 14 and 54 weeks ((Simple Endoscopic Score for CD (SES-CD)≤2(the higher the score, the more severe the disease, heavy activity (SES-CD): >15 points) )
Mucosal healing of different treatment regimens | 14 and 54 weeks
  Mucosal healing rate at 14 and 54 weeks ((Simple Endoscopic Score for CD (SES-CD)=0 (the higher the score, the more severe the disease, heavy activity (SES-CD): >15 points) );
C-reactive protein of different treatment regimens | 14 and 54 weeks
  Changes of serum C-reactive protein from baseline at 14 and 54 weeks;
Erythrocyte sedimentation rate of different treatment regimens | 14 and 54 weeks
  Changes of serum erythrocyte sedimentation rate from baseline at 14 and 54 weeks;
Fecal calprotectin of different treatment regimens | 14 and 54 weeks
  Changes of serum fecal calprotectin from baseline at 14 and 54 weeks;
Intestinal flora of different treatment regimens | 14 and 54 weeks
  Changes in intestinal flora from baseline at 14 and 54 weeks; Fecal 16S rDNA or metagenome sequencing was performed. Fecal samples were obtained from donor and recipient. The fecal samples and isolated microbiota samples were frozen immediately and underwent DNA extraction using standard methods

OTHER OUTCOMES:
Effectiveness and safety | 102 weeks
  Record the incidence of adverse events/adverse reactions (observed at 102 weeks) after the first dose, accurately and specifically describe the incidence of adverse events (such as abdominal pain, fever, allergies, bloating, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Zhihua Huang Huang, Pro, Study Director — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Wuhan, 430030, Wuhan, China

IPD SHARING:
Plan to Share IPD: Yes
The Study Protocol has been uploaded ClinicalTrials.gov
Supporting Information: Study Protocol
Time Frame: 2024.10-2026.10
Access Criteria: Ipds can only be shared with the consent of the principal investigator

REFERENCES:
- See also: Mainly the incidence of IBD — https://pm.yuntsg.com/details.html?pmid=29050646&key=Ng%20SC,%20Shi%20HY,%20Hamidi%20N,%20et%20al.%20worldwide%20incidence%20and%20prevalence%20of%20inflammatory%20bowel%20disease%20in%20the%2021st%20century:%20a%20systematic%20review%20of%20population-based%20studies.%20Lancet.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/34/NCT06673134/Prot_SAP_000.pdf